CLINICAL TRIAL: NCT00093548
Title: A Phase I/II Trial Testing Immunization With AFP + GM-CSF Plasmid Prime And AFP Adenoviral Vector Boost In Patients With Hepatocellular Carcinoma (AFP Prime-Boost Protocol)
Brief Title: Vaccine Therapy in Treating Patients With Stage II, Stage IIIA, Stage IIIB, or Stage IVA Liver Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000389221; UCLA-0302008-02
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized resectable adult primary liver cancer; localized unresectable adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

INTERVENTIONS:
Biological: alpha fetoprotein adenoviral vector vaccine
Biological: alpha fetoprotein plasmid DNA vaccine
Biological: sargramostim plasmid DNA hepatocellular carcinoma vaccine adjuvant

SUMMARY:
RATIONALE: Vaccines made from DNA and a gene-modified virus may make the body build an immune response to kill tumor cells. Giving booster vaccinations may make a stronger immune response and prevent or delay the recurrence of liver cancer.

PURPOSE: This phase I/II trial is studying the side effects and best dose of vaccine therapy and to see how well it works in treating patients with stage II, stage IIIA, stage IIIB, or stage IVA liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and maximum tolerated dose of adjuvant vaccination comprising alpha fetoprotein (AFP) plasmid DNA and sargramostim (GM-CSF) plasmid DNA followed by AFP adenoviral vector boost in patients with HLA-A*0201-expressing stage II-IVA hepatocellular carcinoma.

Secondary

* Determine the optimal biological dose of this regimen, as defined by the generation of AFP-specific immunity, in these patients.
* Determine disease-free survival of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of alpha fetoprotein (AFP) adenoviral vector boost.

Patients receive vaccination comprising AFP plasmid DNA and sargramostim (GM-CSF) plasmid DNA intramuscularly (IM) on days 1, 30, and 60 in the absence of unacceptable toxicity. Patients then receive boost immunization comprising AFP adenoviral vector IM and intradermally on day 90.

Cohorts of 3-6 patients receive escalating doses of AFP adenoviral vector boost until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed monthly for 3 months and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 3-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatocellular carcinoma

  * Stage II-IVA disease

    * No active disease after local or regional therapy (e.g., surgical resection, radiofrequency ablation, cryoablation, or ethanol injection)
* Serum alpha fetoprotein > upper limit of normal
* HLA-A*0201 positive by DNA subtyping

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin > 9.0 g/dL (transfusion independent)
* Platelet count > 50,000/mm^3
* Absolute neutrophil count > 1,000/mm^3

Hepatic

* Child Pugh class A or B liver function
* Hepatitis B or C viral infection allowed

Renal

* Not specified

Cardiovascular

* No New York Heart Association class III or IV cardiac insufficiency
* No coronary artery disease

Immunologic

* HIV negative
* No other acute viral, bacterial, or fungal infection requiring therapy
* No allergy to study agents
* No history of opportunistic infection
* No high serum titer of neutralizing anti-adenoviral antibodies
* No congenital or acquired condition resulting in an inability to generate an immune response

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective double-method (including a barrier method) contraception
* No other condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 30 days since prior chemotherapy
* No concurrent cytotoxic chemotherapy

Endocrine therapy

* At least 30 days since prior steroid therapy
* No concurrent steroid therapy, including corticosteroids

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* No prior organ allograft

Other

* At least 2 weeks since prior therapy for acute infection
* No concurrent immunosuppressive therapy
* No concurrent cyclosporine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, MD, Study Chair — Jonsson Comprehensive Cancer Center

REFERENCES:
- [Derived] Butterfield LH, Economou JS, Gamblin TC, Geller DA. Alpha fetoprotein DNA prime and adenovirus boost immunization of two hepatocellular cancer patients. J Transl Med. 2014 Apr 5;12:86. doi: 10.1186/1479-5876-12-86. PMID 24708667